CLINICAL TRIAL: NCT05310045
Title: Prevention of Modifiable Cancer Risks in Informal Caregivers of Cancer Patients: Implementation and Evaluation of a Personalised Intervention for Vulnerable Informal Caregivers at Increased Risk of Cancer
Brief Title: Personalised Primary Prevention Intervention for Vulnerable Informal Caregivers at Increased Risk of Cancer
Acronym: PREV-AIDANT
Status: Completed | Type: Observational
Sponsor: Centre Leon Berard (Other)
Responsible Party: Sponsor
Other Study IDs: PREV-AIDANT
Record Dates: First submitted 2022-03-16; First posted 2022-04-04 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2025-03

CONDITIONS: Informal Caregivers; Healthy Volunteers; Family; Spouses
Keywords: primary prevention; informal caregivers; cancer risk; personalised intervention

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Behavioral: Personalised primary prevention intervention — Personalised primary prevention intervention
  1. Consultation 1
     * Assess caregiver's situation regarding their cancer risk factors
     * Explain the causal links between risk factors and cancer
     * Inform about national recommendations to prevent and limit cancer risk
     * Clarify informal caregiver situation with respect to national screening programs
     * Define a personalised primary prevention program
  2. Implementation: personalised primary prevention program
     * Carried out by the informal caregiver
     * Supervised by the coordinating nurse
  3. Consultation 2
     * Assess prevention actions realised by informal caregiver in relation to actions defined in the personalised primary prevention program
     * Identify barriers and facilitators to their implementation whether actions or no actions have been done.
     * Adapt the personalised primary prevention program to informal caregiver needs.

SUMMARY:
Today, 40% of cancers are linked to modifiable risk factors and could thus be preventable. Primary prevention, which allows individuals to be informed and aware of health recommendations and possible actions before the onset of a cancer, is thus a major public health issue.

Around 11 million of French citizens are informal caregivers, i.e. people who regularly and frequently provide a non-professional help to do all or part of daily life activities for a dependent person with a disability, disease, or due to age. In cancer, there are around 5 million of informal caregivers in France.

Studies have shown that informal caregivers of cancer patients are not only at risk for stress, anxiety, poor health, diminished quality of life, but also that they adopt so-called "risk behaviours" (e.g., increased smoking or alcohol consumption, unbalanced eating habits rich in fat, sugar and ultra-processed foods, sedentary lifestyle, etc.). These behaviours may develop or worsen co-morbidities and/or promote cancer development, outside hereditary context. Moreover, for certain types of cancer, related and unrelated family caregivers have a higher risk of developing cancer because they share the same lifestyle including the same risk factors. However, compared to general population, informal caregivers of cancer patients, have an increased risk perception and motivation to change a so-called unhealthy lifestyle.

In this context, our goal is to test the feasibility and acceptability of a personalised primary prevention intervention designed to informal caregivers of cancer patients at increased risk of cancer.

The intervention will be first designed to first-degree relatives and partners/spouses of a patient treated at Léon Bérard Center.

Developed in the Léon Bérard comprehensive cancer centre in close relation with outpatient care and based on an informal caregiver's tracking questionnaire, the intervention will be composed of two consultations with a physician trained in primary prevention and information and referral to health prevention structures.

As primary objectives, acceptability will be assessed based on informal caregivers' satisfaction and feasibility based on their participation rates.

As secondary objectives, informal caregivers' knowledge and risk perception will be assessed based on questionnaires and intention to change or change behaviour will be noted and analysed through individual semi-structured interviews.

ELIGIBILITY:
Inclusion Criteria:

* First-degree relative and partner/spouse of a patient treated at the Centre Léon Bérard;
* At increased risk of cancer
* Aged between 18 and 75 years;
* No diagnosis of genetic predisposition to cancer and no personal or informal history suggesting genetic predisposition;
* Able to complete a questionnaire in French, alone or with the help of a relative (persons with visual, mute, motor, hearing or intellectual disabilities will be included as long as they are able to complete a questionnaire alone or with the help of a relative);
* Being informed and not opposed to the study ;
* Having completed the entire tracking questionnaire and wishing to be contacted.

Exclusion Criteria:

* Related or unrelated relative not considered as an informal caregiver for the patient;
* Minor informal caregiver;
* Informal caregiver with a history of cancer;
* Patient under care at the Institute of Hematology and Pediatric Oncology;
* Individuals of legal age protected by law.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: First-degree relative and partner/spouse of a patient treated at the Centre Léon Bérard, at increased risk of cancer
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2022-04-04 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-15 (Actual)

PRIMARY OUTCOMES:
Acceptability of the intervention | At the end of the personalised primary prevention intervention (4 to 6 months after inclusion)
  Acceptability will be assessed based on informal caregivers' satisfaction.
Feasibility of the intervention | At the end of the personalised primary prevention intervention (4 to 6 months after inclusion)
  Feasibility will be assessed based on informal caregivers' participation rates.

SECONDARY OUTCOMES:
Adherence of informal caregivers to the different stages of the study: filling in the questionnaire | At the pre-inclusion
  Informal caregivers are identified with a tracking questionnaire. The percentage of informal caregivers who responded to the tracking questionnaire will be measured.
Adherence of informal caregivers to the different stages of the study: attendance to consultations | At the end of the 1st (2 to 6 weeks after inclusion) and the 2nd consultation (4 to 6 months after inclusion)
  The personalised primary prevention intervention is composed of 2 consultations. The percentage of informal caregivers who participated to the 1st and 2nd consultation will be measured.
Experience, of informal caregivers who have benefited from all the personalised primary prevention intervention | After the 2nd consultation (4 to 6 months after inclusion)
  Experience will be analysed using individual semi-structured interviews.
Short-term impact of the personalised primary prevention intervention: knowledge | Before the 1st (2 to 6 weeks after inclusion) and the 2nd consultation (4 to 6 months after inclusion)
  Knowledge will be measured by informal caregiver's through a knowledge score based on a questionnaire.
Short-term impact of the personalised primary prevention intervention: cancer risk perception | Before the 1st (2 to 6 weeks after inclusion) and the 2nd consultation (4 to 6 months after inclusion)
  Cancer risk perception will be measured by informal caregiver's through a cancer risk perception score, based on a questionnaire.
Short-term impact of the personalised primary prevention intervention: Intention/behaviour change | During the second consultation (4 to 6 months after inclusion)
  Intention/behaviour change will be measured by the percentage of actions planned in the personalised primary prevention programme and actually carried out by the informal caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: Béatrice FERVERS, Principal Investigator — Centre Léon Bérard (CLB)
Locations (1):
- Centre Leon Berard, Lyon, France

IPD SHARING:
Plan to Share IPD: No
We are not planning to share IPD